CLINICAL TRIAL: NCT02131558
Title: The Feasibility and Benefits of Using Indocyanine Green and Near-infrared Fluorescence Imaging to Detect Sentinel Lymph Nodes in Patients With Endometrial Cancer
Brief Title: Indocyanine Green and Near-infrared Fluorescence Imaging to Detect Sentinel Lymph Nodes in Patients With Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Valena Wright, Director of Minimally Invasive Gynecologic Surgery, Lahey Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-017
Record Dates: First submitted 2014-04-07; First posted 2014-05-06 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Endometrial Cancer; Sentinel Lymph Node Detection
Keywords: Endometrial cancer; Sentinel lymph node; Indocyanine green; Near infrared imaging
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICG Dye (Experimental): Patients received injections of Indocyanine green (ICG) for sentinel lymph node (SLN) visualization using near-infrared (NIR) imaging.
  Interventions: Procedure: ICG Dye

INTERVENTIONS:
Procedure: ICG Dye — ICG Dye injections

SUMMARY:
Patients with endometrial cancer who have planned robotic laparoscopic hysterectomy and full bilateral pelvic and para-aortic lymphadenectomy will receive injections of a fluorescent dye, Indocyanine green (ICG). ICG spreads through the lymphatic system, and will be visualized using near-infrared (NIR) imagers. Upon visualization of the path of the ICG, sentinel lymph nodes (SLNs), the first nodes to receive drainage from the primary tumor, will be identified. SLNs will be surgically removed and provided to Pathology for evaluation. Non-sentinel nodes will also be surgically removed, as is consistent with routine medical care for these patients, and given to Pathology for evaluation. A positive SLN may be the most accurate identifier of the extra-uterine spread of disease, and will provide information about the extent of surgical node removal necessary.

ELIGIBILITY:
Inclusion Criteria:

* Adult women patients (>18 years of age and <90 years of age)
* Research authorization (consent)
* Pre-operative diagnosis of clinical Stage 1 endometrial cancer
* Pre-operative indications of grade 3 tumor, and/or tumor size greater than 2 cm in size
* Scheduled and consented to undergo robotic hysterectomy and surgical staging, including bilateral pelvic and para-aortic lymphadenectomy

Exclusion Criteria:

* Severe coagulopathy or severe thrombocytopenia
* Severe anemia
* Severe cardio-pulmonary comorbidities demanding minimization of operative time
* History of liver disease
* Iodide allergy
* Emergent operation
* Additional surgical risk as determined during surgery at the discretion of the attending
* Impaired capacity to make informed medical decisions

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05; Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
Detection of sentinel lymph node(s) | Detection of SLNs will occur within surgery, on average this surgery will take "1-2 hours" for each participant
  The primary outcome is to determine whether sentinel lymph nodes (SLN) were accurately visualized using Indocyanine green (ICG) and near-infrared (NIR) imaging.

SECONDARY OUTCOMES:
Comparison between sentinel node status for disease and non-sentinel node disease status | Following surgery and pathological evaluation of all removed nodes, up to "1 year"
  The pathological evaluation of the sentinel lymph nodes (positive or negative) will be compared to the status of the non-sentinel nodes removed to determine whether the sentinel nodes accurately reflected the same status as the non-sentinel nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Valena Wright, MD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States

REFERENCES:
- [Background] Rossi EC, Jackson A, Ivanova A, Boggess JF. Detection of sentinel nodes for endometrial cancer with robotic assisted fluorescence imaging: cervical versus hysteroscopic injection. Int J Gynecol Cancer. 2013 Nov;23(9):1704-11. doi: 10.1097/IGC.0b013e3182a616f6. PMID 24177256
- [Background] Rossi EC, Ivanova A, Boggess JF. Robotically assisted fluorescence-guided lymph node mapping with ICG for gynecologic malignancies: a feasibility study. Gynecol Oncol. 2012 Jan;124(1):78-82. doi: 10.1016/j.ygyno.2011.09.025. Epub 2011 Oct 11. PMID 21996262
- [Background] Abu-Rustum NR. Update on sentinel node mapping in uterine cancer: 10-year experience at Memorial Sloan-Kettering Cancer Center. J Obstet Gynaecol Res. 2014 Feb;40(2):327-34. doi: 10.1111/jog.12227. PMID 24620369
- [Background] Abu-Rustum NR. Sentinel lymph node mapping for endometrial cancer: a modern approach to surgical staging. J Natl Compr Canc Netw. 2014 Feb;12(2):288-97. doi: 10.6004/jnccn.2014.0026. PMID 24586087